CLINICAL TRIAL: NCT03357068
Title: Effect of Citric Acid Demineralization on Autogenous Bone Blocks Consolidation in Humans: Qualitative, Quantitative and Immunohistochemical Analysis
Brief Title: Effect of Citric Acid Demineralization on Autogenous Bone Blocks Consolidation in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Carla Andreotti Damante, Associate professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FOBblock
Record Dates: First submitted 2017-11-22; First posted 2017-11-29 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Alveolar Bone Atrophy; Bone Resorption
MeSH Terms: conditions — Alveolar Bone Loss; Bone Resorption | interventions — Acids

STUDY DESIGN:
Intervention Model Description: Split mouth design - one side of mouth is test group, other side is control group
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Autogenous bone block surgery without treatment of bone surfaces.
  Interventions: Procedure: Control
- Acid (Experimental): Autogenous bone block surgery with citric acid treatment of bone block and recipient site
  Interventions: Procedure: Acid

INTERVENTIONS:
Procedure: Control — Control side will receive only perforations on recipient site, which is the conventional technique for bone blocks graft.
  Arms: Control
Procedure: Acid — Test side will receive treatment with citric acid (10%) for 30s at bone block surface and recipient site
  Arms: Acid

SUMMARY:
This study evaluates the effect of citric acid demineralization in autogenous bone blocks consolidation. Half of participants will receive citric acid treatment at the bone block and recipient site. Other half will receive no demineralization treatment.

DETAILED DESCRIPTION:
Autogenous bone grafts are indicated in areas where there is not enough bone height and/or width for implant installation. Treatment of bone surfaces with citric acid, promote a slight demineralization on surface that mimic natural processes of bone demineralization by osteoclasts. Thus, this treatment could accelerate the process of autogenous bone block consolidation to its recipient site.

ELIGIBILITY:
Inclusion Criteria:

* Presence of atrophic anterior maxilla (width 1.5 to 4 mm)
* Absence of active periodontal disease.
* Enough bone width on donor sites (oblique line or ment)

Exclusion Criteria:

* Systemic disease that impede surgical procedure as blood diseases, endocrine diseases, impaired coagulation
* Smokers
* Pregnant women
* Patients receiving radiotherapy or chemotherapy
* Patients using bisphosphonates

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-12-22 (Actual)

PRIMARY OUTCOMES:
Clinical bone block consolidation | 5 months
  Absence of fibrous tissue by clinical observation
Computerized tomography images bone block consolidation | 5 months
  Absence of images compatible to fibrosis in cone beam computerized tomography images
Histological bone block consolidation | 5 months
  Absence of fibrous tissue between bone block and recipient site in histological images.

SECONDARY OUTCOMES:
Bone width | 5 months
  Measurement of bone width in mm on cone beam computerized tomography. Ideal if >6 mm.

CONTACTS AND LOCATIONS:
Locations (1):
- Bauru School of Dentistry, Bauru, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rezende ML, Consolaro A, Sant'Ana AC, Damante CA, Greghi SL, Passanezi E. Demineralization of the contacting surfaces in autologous onlay bone grafts improves bone formation and bone consolidation. J Periodontol. 2014 May;85(5):e121-9. doi: 10.1902/jop.2013.130298. Epub 2013 Oct 30. PMID 24171500